CLINICAL TRIAL: NCT00259441
Title: Prevention of Radiocontrast Media Induced Nephropathy by Short-Term High-Dose Statin in Renal Insufficiency Undergoing Coronary Angiography (PROMISS)
Brief Title: PROMISS: Simvastatin Prevents the Contrast Induced Acute Renal Failure in Patients With Renal Insufficiency Undergoing Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-0509-517-158
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Kidney Failure
Keywords: Kidney failure; Contrast media; Prevention; Simvastatin
MeSH Terms: conditions — Renal Insufficiency | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
The contrast induced kidney toxicity has been known to affect the mortality and morbidity in the patients undergoing coronary angiography. But the mechanism and therapeutic strategy for it is not well known. Nowadays, it is reported that the N-acetylcysteine may have preventive effects for contrast induced kidney toxicity with its antioxidant effects.The statins have been reported to have many other effects other than the lipid lowering effect-including antioxidant effect, so we hypothesized that the antioxidant effect of simvastatin may prevent the contrast induced kidney toxicity.

DETAILED DESCRIPTION:
The simvastatin may prevent the contrast agent induced acute renal failure in the patients with underlying renal insufficiency who is undergoing the coronary angiography. The effect may derive from the antioxidant function of simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Angina patients
* Patients who is required the coronary catheterization
* creatinine clearance rates ≤60 mL/min using the Cockcroft-Gault formula Patients who undergo coronary catheterization
* Age of 19 or over 19

Exclusion Criteria:

* pregnancy
* lactation
* having received contrast media within 7 days of study entry
* emergent coronary angiography
* acute renal failure
* end-stage renal disease requiring dialysis
* history of hypersensitivity reaction to contrast media
* cardiogenic shock
* pulmonary edema
* multiple myeloma
* mechanical ventilation
* parenteral use of diuretics
* use of N-acetylcysteine
* use of metformin or nonsteroidal anti-inflammatory drugs within 48 hours of the procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2005-02; Study Completion 2006-03

PRIMARY OUTCOMES:
The mean peak increase of serum creatinine concentration during day1 and day2.

SECONDARY OUTCOMES:
Incidence of contrast induced nephropathy, defined as either a relative increase in serum creatinine from baseline of >=25% or an absolute increase of >=0.5mg/dL(44.2µmol/L) during days 1 and 2.
Proportion of patients exhibiting an increase in serum creatinine of >=0.5mg/dL(44.2µmol/L), the proportion with a >=1.0 mg/dL(88.4µmol/L) increase in serum creatinine, and the mean peak increase in serum creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, M.D., Ph.D., Study Chair — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center; Hyo-Soo Kim, M.D.,Ph.D., Study Director — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center; Sang-Ho Jo, M.D., Principal Investigator — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center; Bon-Kwon Koo, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center
Locations (1):
- Seoul National University Hospital , Cardiovascular Center, Seoul, South Korea

REFERENCES:
- [Derived] Jo SH, Koo BK, Park JS, Kang HJ, Cho YS, Kim YJ, Youn TJ, Chung WY, Chae IH, Choi DJ, Sohn DW, Oh BH, Park YB, Choi YS, Kim HS. Prevention of radiocontrast medium-induced nephropathy using short-term high-dose simvastatin in patients with renal insufficiency undergoing coronary angiography (PROMISS) trial--a randomized controlled study. Am Heart J. 2008 Mar;155(3):499.e1-8. doi: 10.1016/j.ahj.2007.11.042. Epub 2008 Jan 30. PMID 18294484